CLINICAL TRIAL: NCT06429423
Title: Acute Psychological and Physiological Exercise Effects Among Patients With Stress-related Exhaustion Disorder. Role of Exercise Intensity.
Brief Title: Effects of Acute Physical Activity in Patients With Exhaustion Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victoria Blom (Other)
Collaborators: Avonova Health AB (Unknown); Jenny Kling, Doctoral student, licensed psychologist, The Swedish School of Sport and Health Sciences (Unknown)
Responsible Party: Sponsor-Investigator, Victoria Blom, Associate professor in psychology, head of department Institution for physical activity and health, licensed psychologist, The Swedish School of Sport and Health Sciences
Organization: The Swedish School of Sport and Health Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-04943-01
Record Dates: First submitted 2024-02-06; First posted 2024-05-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Exhaustion; Syndrome
Keywords: burnout; fatigue; psychological stress; physical activity; acute exercise; mood; heart rate variability
MeSH Terms: conditions — Syndrome; Burnout, Psychological; Fatigue; Stress, Psychological; Motor Activity

STUDY DESIGN:
Intervention Model Description: The design is a two-armed intervention with two groups (30+30), one which is patients with ED, and the other an age- and sex matched control group with overall healthy individuals. The two trial conditions will be performed in a counter-balanced randomized order on two separate days with at least one week apart. Participants will be randomized regarding order of two different intensities of physical activity bouts. The participants will perform the two conditions of physical activity bouts at approximately the same time in the morning/forenoon with at least 1 week in between conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exhaustion disorder (ED) (Experimental): Patients with diagnosed exhaustion disorder (F43.8A in Swedish ICD-10).
  Interventions: Behavioral: Acute exercise low intensity; Behavioral: Acute exercise moderate intensity
- Control group (Active Comparator): Age- and sex-matched healthy control participants.
  Interventions: Behavioral: Acute exercise low intensity; Behavioral: Acute exercise moderate intensity

INTERVENTIONS:
Behavioral: Acute exercise low intensity — A 15-minute exercise on low intensity on a cycle ergometer. Immediately before, immediately after and 30 minutes after exercise participants will fill out questionnaires regarding feelings of fatigue, energy, anxiety and stress and measure saliva cortisol. Three times during the exercise, they will rate level of exertion (RPE) and feelings of distress on a VAS-scale.
  During the 24 hours following the exercise bout they will wear a heart rate strap and an accelerometer measuring heart rate variability and activity level. Twice during that time, once in the evening, and once in the morning after, participants will answer questionnaires regarding mood state.
Behavioral: Acute exercise moderate intensity — A 15-minute exercise on moderate intensity on a cycle ergometer. Immediately before, immediately after and 30 minutes after exercise participants will fill out questionnaires regarding feelings of fatigue, energy, anxiety and stress and measure saliva cortisol. Three times during the exercise, they will rate level of exertion (RPE) and feelings of distress on a VAS-scale.
  During the 24 hours following the exercise bout they will wear a heart rate strap and an accelerometer measuring heart rate variability and activity level. Twice during that time, once in the evening, and once in the morning after, participants will answer questionnaires regarding mood state.

SUMMARY:
A new stress-related diagnosis, Exhaustion disorder (ED), was introduced in the Swedish version of ICD-10 in 2005 and has since then increased rapidly. The condition is long-lasting and debilitating, characterized by considerable and persistent fatigue, insomnia, and impaired cognitive function. The diagnosis is still relatively unexplored and there is no consistent knowledge of, among other things, which interventions that work. Research indicates that physical activity can have positive effects on depression, anxiety, and stress. However, there is little knowledge today about the relationship between the dose of physical activity and stress-related illness. It is also not clear how physical activity can be used in the treatment of stress-related illness. The purpose of this project is to gain increased knowledge about the immediate physiological and psychological effects of physical activity for people with diagnosed ED. The project will investigate the psychological and physiological effects of two different intensities of physical activity in people with ED compared to healthy controls. The information from the study also aims to provide a basis for a second part of the project where treatment including physical activity is carried out with people with ED, in a randomized controlled design.

DETAILED DESCRIPTION:
Background A new stress-related diagnosis, exhaustion disorder (ED), was introduced in the Swedish version of ICD-10 in 2005, and has since then increased rapidly. The condition is long-lasting and debilitating, characterized by considerable and persistent fatigue, insomnia and impaired cognitive function. The diagnosis is still relatively unexplored and there is no consistent knowledge of, among other things, which interventions that work.

There is extensive research on the association between mental health and physical activity in general and exercise specifically. When it comes to long-term, or habitual, exercise, it is established that it has beneficial effects on different aspects of mental health and physical activity interventions are helpful for people with mental illness. The most widely studied mental health-issues are depression, anxiety, and stress, and a recent umbrella review concludes that habitual exercise is beneficial for symptom reduction for depression, anxiety, and stress across different populations. Epidemiological evidence shows that physical activity is associated with lowered risk of experiencing fatigue and reduced energy.

Little is known about how physical activity in general and more specifically different intensities of physical activity affects people with ED. Does it have adverse effects or is it beneficial? This is imperative when it comes to intervention- and treatment planning for these patients. No studies have been done specifically on ED before with this focus. Although an acute study cannot show the optimal physical activity program, it can give insight into the relation between between ED and exercise. This in turn can help us construct better designs of exercise programs for this patient group.

Research aims and questions The purpose of the study is to gain increased understanding of the psychological and physiological response to acute exercise in ED-patients compared to a healthy population, and to determine if that response differs between two different intensities of exercise (low and moderate). The focus is on transient emotional states and how they might fluctuate in response to exercise. Specifically subjective feelings of fatigue, energy, anxiety, psychological discomfort, perceived exertion, recovery, and stress is studied. Salivary cortisol and heart rate variability (HRV) are the biomarkers in focus.

Knowledge from the study is planned to be used in the designing of a physical activity program as part of a treatment program for ED. The design can give us information about whether short bouts of exercise can have mood-altering effects in this patient group, and auonomic reactivity to physical activity.

Research questions:

1. Does level of fatigue, vigor/energy, state anxiety, and perceived stress differ between groups (ED/controls) and/or between exercise intensities (mild/moderate) and/or between timepoints (pre/post/30minpost/6hpost/24hpost)?
2. Does the level of subjective discomfort and perceived exertion differ between groups (ED/controls) and/or between exercise intensities (mild/moderate) and/or between time points (pre/5min/10min/15min)?
3. Does the level of salivary cortisol differ between groups (ED/controls) and/or between exercise intensities (mild/moderate) and/or between time points (pre/post/30 min post)?
4. Does level of heart rate variability (HRV) differ between groups (ED/controls) and/or between exercise intensities (mild/moderate) and/or between timepoints (pre/post/30minpost/6hpost/24hpost)?

If significant differences are found, intercation effects between the different variables will also be studied, as well as potential moderating variables.

Methods Study design The design is a two-armed trial (low and moderate intensity of physical activity) with two groups, one which is patients with ED, and the other an age- and sex matched control group with overall healthy individuals, that include sequential assessments of fatigue and energy states, stress, perceived exertion, perceived psychological distress and state anxiety.

Participants Approximately 30 patients with diagnosed exhaustion disorder (F43.8A in ICD-10-SE) and 30 age- and sex-matched healthy control participants are recruited for the study. ED-patients are recruited through occupational health care Avonova and through advertisement in social media Facebook and Instagram. Inclusion criteria in the studies for ED-patients: confirmed primary diagnosis ED by a physician; assessed to not be in the acute phase of ED; age of 35-55 years; considered by a physician and/or a psychologist as suitable for participating in a study including performing physical activity. Healthy control participants are recruited via the same social media channels as ED-patients. Inclusion criteria: age of 35-55 years; self-reported good health (no known somatic or psychiatric disease); considered as suitable for participating in a study including performing physical activity. Mini International Neuropsychiatric Interview 6.0.0. (MINI), as well as an additional diagnostic questionnaire targeting stress-related disorders based on diagnostic criteria from ICD-11, will be conducted with both ED-patients and healthy controls, to ensure the inclusion- and exclusion criteria. MINI is a diagnostic interview for the major DSM-IV psychiatric disorders. The participants will receive thorough written information about the study and written informed consent will be obtained before inclusion. The study was approved by the Regional Ethical Review Board in Linköping, Sweden (Approval Nr. 2022-04943-01) and will be conducted in accordance with the ethical principles of the Declaration of Helsinki.

Procedure The study takes place in a laboratory setting at GIH on three different days, separated by at least one week. Before enrollment, participants complete an online administered screening questionnaire measuring exhaustion, burnout, and diagnostic and general health information. Eligible participants are invited to GIH for a familiarization visit, where a structured clinical interview (MINI and stress diagnoses questionnaire) is performed. Participants will also complete a submaximal cardiorespiratory fitness test (CRF) to estimate maximal aerobic capacity. The test is performed on a calibrated mechanically braked cycle ergometer (model 828E, Monark, Varberg, Sweden) for 8 min. Pedal frequency throughout the test is 60 rpm. Cycling resistance starts at 0,5 kilopond (kp) for 4 minutes and is increased to a personalized higher work rate, which lasts for 4 minutes. VO2max is estimated from these 8 minutes using heart rate data collected during the test. The result on this test will be used in determining each participant's correct intensity level on the two trial conditions.

Conditions The two trial conditions are performed in a counter-balanced and randomly assigned order. The participants perform the two conditions of physical activity bouts at approximately the same time in the morning/forenoon (start time of test visit is either 8:30 or 10:30 a.m.) with at least one week in between conditions. The participants have the same test start time at the two test visits. At each test session participants perform a 22-minute exercise on a cycle ergometer (model 839E, Monark, Varberg, Sweden). Immediately before and at three time points during the exercise (after 5, 10, and 15 minutes on the low or moderate intensity), they rate level of exertion (RPE) and feelings of psychological distress on a VAS-scale. Immediately before, immediately after, 30 minutes after, 6 hours after, and 24 hours after exercise participants fill out questionnaires regarding feelings of fatigue, energy, anxiety, recovery, and stress. Participants wear a H10 heart rate sensor and Vantage M2 monitor (Polar, Kempele, Finland) for a little more than 24 hours, starting approximately 30 minutes before the exercise. HRV parameters will be calculated from 5-min window recordings using the software Kubios HRV (University of Eastern Finland, Kuopio, Finland), immediately before (pre), immediately after (post), 30 minutes after (30 min post), 6 hours after (6h post), and 24 hours after (24h post) exercise. Since HRV is influenced by several factors (caffeine intake, alcohol consumption, circadian rhythm, stress (both mental and physical), exercise, food- and water intake, certain medications, bladder filling, respiratory rate, and posture) these factors will be controlled for when at GIH. Salivary cortisol is collected pre, post and 30 min post exercise using Sarstedt Salivette Cortisol (Sarstedt, Nümbrecht, Germany). The follow-up measurements will determine the trajectory of the cortisol and HRV post-exercise. During the 24 hours following the exercise bout physical activity pattern is measured using a hip-worn accelerometer (Actigraph GT3X). Accelerometer data will be processed in Actilife.

There are two experimental exercise conditions, where participants will exercise at two different intensity levels. The intensity levels are standardized across participants by using results from EKBLOM-BAK test to determine a low and moderate intensity. Low intensity is defined as 40% and moderate intensity is defined as 55% of the participant's individual estimated VO2max. The 22-minute exercise starts with a 6-minute warm-up, with a load increase after 1 and 3 minutes and lowered load at the last minute. Then follows a 15-minute bout on either low or moderate intensity, that ends with a 1-minute cool-down. One of the researchers will be present during the complete test to assure correct intensity and length.

Baseline measures

In the week before the familiarization visit each participant completes a digitally administered questionnaire that includes socio-demographic and general health information together with the following questionnaires:

* Exhaustion disorder. Karolinska Exhaustion Disorder Scale (KEDS) was developed for the assessment of ED symptoms. It consists of nine items with a scale range of 0-54 and a cut-off of 19 has been proposed in the discrimination between healthy subjects and patients with ED.
* Burnout. Shirom-Melamed Burnout Questionnaire/Measure (SMBQ/SMBM) is widely used in measuring burnout. SMBM-12 is a short version with twelve items which captures core concepts of burnout: emotional and physiological exhaustion (e.g., "I feel tired"), and cognitive weariness (e.g., "I feel I am not thinking clearly"). A global score of burnout is calculated. SMBM-12 has good composite reliability and convergent validity.
* Trait anxiety. The trait subscale of The State-Trait Anxiety Inventory (STAI). Respondents rate how they generally feel on a 4-point Likert Scale (e.g., "I feel nervous and rested"). A global score of a general and enduring trait anxiety is calculated.
* Depression. Patient Health Questionnaire (PHQ-9) measures depression in line with DSM-IV. Respondents rate depression symptoms the last two weeks on a 4-point Likert Scale (e.g., "Little interest or pleasure in doing things").
* Sleep. Pittsburgh Sleep Quality Index (PSQI) is widely used in measuring sleep quality. It consists of 19 items that form seven components of retrospective sleep quality (1 month) and a global score.
* Physical activity. Saltin-Grimby Physical Activity Level Scale (SGPALS) is a four-level single-item instrument which has acceptable validity for measuring level of physical activity.
* Exercise attitudes. Two subscales of the Exercise Benefits/Barriers Scale (EBBS) were included: Psychological Outlook Subscale (benefits), and Physical Exertion Subscale (barriers).

2-3 days after the familiarization visit, heart rate variability (HRV) and physical activity pattern is measured during a 24-hour baseline measurement. Participants get oral and written instructions on the familiarization visit on how to initialize and conduct this measurement with a H10 heart rate sensor and Vantage M2 monitor together with a hip-worn accelerometer (Actigraph GT3X). Twice during the 24h-measurement, digital questionnaires including Single Item stress Question (SISQ), the vigor and fatigue subscales of Profile of Mood States (POMS), single-item recovery question, and state subscale of The State-Trait Anxiety Inventory (STAI-Y1) are completed.

Data analysis For each of the psychological variables (perceived exertion, psychological discomfort, fatigue, energy/vigor, state anxiety, and stress) a three factorial (group, time, intensity) ANOVA with repeated measures design will be the first hand choice if parametric assumptions are met. A secondary stratified analysis will be performed exploring potential variables that influenced the primary and secondary psychological variables.

For the data analysis of physiological variables, data analysis are yet to be decided. This will be done though before looking at the data.

ELIGIBILITY:
Inclusion Criteria:

For ED-patients:

* Confirmed primary diagnosis ED by a physician
* Assessed to not be in the acute phase of ED
* considered by a physician and/or a psychologist as suitable for participating in a study including performing physical activity
* Age of 35-55 years

For control group:

* Self-reported good health (no known somatic or psychiatric disease)
* Age of 35-55 years

Exclusion Criteria:

* Chronic fatigue syndrome (CFS)
* Post-covid
* Dementia
* Bipolar and/or psychotic disorder
* Current substance abuse
* Fibromyalgia
* Elevated suicide risk
* Medication with beta-blockers

Following exclusion criteria is also used, since it is not suitable to perform the EKBLOM-BAK-test:

* chronic obstructive lung disease
* hypertension/dyslipidemia
* cardiovascular disease

If participant has ongoing infection (such as a cold) on testday, testing is delayed until she/he is recovered.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Fatigue | Fatigue is measured in both conditions at the following time-points: immediately before the exercise bout, immediately after the exercise bout, 30 minutes after the exercise bout, 6 hours after the exercise bout, and 24 hours after the exercise bout.
  Fatigue is defined as "a persistent sense of physical, emotional, and/or cognitive tiredness or exhaustion". Feelings of energy and fatigue is measured with the vigor and fatigue subscales of Profile of Mood States (POMS). It assesses short-term mood states and respondents are instructed to rate how the feel "right now". The total score ranges from 0 to 28 and a higher score means a worse outcome. It is a valid and reliable measure of intensities of fatigue and energy mood states and is recommended to be used in experimental settings to measure short-term intensity of energy and fatigue moods.
Energy/vigor | Energy/vigor is measured in both conditions at the following time-points: immediately before the exercise bout, immediately after the exercise bout, 30 minutes after the exercise bout, 6 hours after the exercise bout, and 24 hours after the exercise bout
  The adopted definition of energy is "an individual's potential to perform mental and physical activity". Feelings of energy and fatigue is measured with the vigor and fatigue subscales of Profile of Mood States (POMS). It assesses short-term mood states and respondents are instructed to rate how the feel "right now". The total score ranges from 0 to 32 and a higher score means a better outcome. It is a valid and reliable measure of intensities of fatigue and energy mood states and is recommended to be used in experimental settings to measure short-term intensity of energy and fatigue moods.
State anxiety | State anxiety is measured in both conditions at the following time-points: immediately before the exercise bout, immediately after the exercise bout, 30 minutes after the exercise bout, 6 hours after the exercise bout, and 24 hours after the exercise bou
  State anxiety will be measured using the 20-item state subscale of The State-Trait Anxiety Inventory (STAI-Y1). Respondents rate how they feel "right now" on a 4-point Likert Scale (e.g., "I am tense"). A global score of the transient condition of state anxiety is calculated, ranging from 20 to 80. Higher scores correlates with greater anxiety. It is extensively used in previous studies of acute exercise and there is support for the STAI-Y1 being sensitive to change in response to acute aerobic exercise.

SECONDARY OUTCOMES:
Stress. | Stress is measured in both conditions at the following time-points: immediately before the exercise bout, immediately after the exercise bout, 30 minutes after the exercise bout, 6 hours after the exercise bout, and 24 hours after the exercise bout.
  To measure subjective stress in the moment the Single Item stress Question (SISQ) was adapted and reformulated to measure stress "right now" instead of "these days". The scale ranges from 1 to 5, and higher scores correlates with higher level of stress.
Perceived psychological discomfort. | SUD is measured in both conditions at the following time-points: immediately before the exercise bout; during the exercise at 3 time points: 5 min into the exercise, 10 min into the exercise, and 15 min into the exercise
  Subjective Units of Distress (SUD) is used to assess the strength of subjective discomfort during the exercise bout. The respondent is asked to rate on a scale from 0 to 10 how much discomfort they experience. The scale ranges from 0 10 and a higher score indicates more discomfort.
Perceived Exertion. | RPE is measured in both conditions at the following time-points: immediately before the exercise bout; during the exercise at 3 time points: 5 min into the exercise, 10 min into the exercise, and 15 min into the exercise
  Borg's 6-20 rating of perceived exertion scale (RPE) was used to assess exertion during exercise. It is a single-item scale ranging from 6 (not strenuous at all) to 20 (maximally strenuous).
Salivary cortisol | Cortisol is measured in both conditions at the following time points: 10 minutes before each exercise bout; 5 minutes after each exercise bout; and 35 minutes after each exercise bout.
  Is used as a biomarker indicator of the HPA-axis response to exercise. Saliva is collected with standard swabs; Sarstedt Salivette Cortisol, then stored and analyzed following standard procedures.
Heart rate variablity (HRV) | HRV is measured in both conditions at the following time points: 5 minutes before exercise bout; ca 8 minutes after exercise bout; and ca 38 minutes after exercise bout.
  Specific measures still to be decided upon. This will be decided before looking at the data.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Blom, Ass. prof., Principal Investigator — The Swedish School of Sport and Health Sciences
Locations (1):
- Victoria Blom, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almén, N., & Jansson, B. (2021). The reliability and factorial validity of different versions of the Shirom-Melamed Burnout Measure/Questionnaire and normative data for a general Swedish sample. International Journal of Stress Management, 28(4), 314-325. https://doi.org/10.1037/str0000235
- [Background] Bjorkman F, Ekblom-Bak E, Ekblom O, Ekblom B. Validity of the revised Ekblom Bak cycle ergometer test in adults. Eur J Appl Physiol. 2016 Sep;116(9):1627-38. doi: 10.1007/s00421-016-3412-0. Epub 2016 Jun 16. PMID 27311582
- [Background] Borg G, Ljunggren G, Ceci R. The increase of perceived exertion, aches and pain in the legs, heart rate and blood lactate during exercise on a bicycle ergometer. Eur J Appl Physiol Occup Physiol. 1985;54(4):343-9. doi: 10.1007/BF02337176. PMID 4065121
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] World Health Organization: The ICD-10 classification of mental and behavioural disorders: Clinical descriptions and diagnostic guidelines. Geneva: World Health Organization, 1992.
- [Background] Lindsater E, Svardman F, Wallert J, Ivanova E, Soderholm A, Fondberg R, Nilsonne G, Cervenka S, Lekander M, Ruck C. Exhaustion disorder: scoping review of research on a recently introduced stress-related diagnosis. BJPsych Open. 2022 Aug 24;8(5):e159. doi: 10.1192/bjo.2022.559. PMID 36458830
- [Background] Singh B, Olds T, Curtis R, Dumuid D, Virgara R, Watson A, Szeto K, O'Connor E, Ferguson T, Eglitis E, Miatke A, Simpson CE, Maher C. Effectiveness of physical activity interventions for improving depression, anxiety and distress: an overview of systematic reviews. Br J Sports Med. 2023 Sep;57(18):1203-1209. doi: 10.1136/bjsports-2022-106195. Epub 2023 Feb 16. PMID 36796860
- [Background] Spielberger, C.D., Gorsuch, R.L., & Lushene, R.E. (1970). The State-Trait Anxiety Inventory: Testmanual. Palo Alto, CA: Consulting Psychologist Press
- [Background] Saltin B, Grimby G. Physiological analysis of middle-aged and old former athletes. Comparison with still active athletes of the same ages. Circulation. 1968 Dec;38(6):1104-15. doi: 10.1161/01.cir.38.6.1104. No abstract available. PMID 5721960
- [Background] Sechrist KR, Walker SN, Pender NJ. Development and psychometric evaluation of the exercise benefits/barriers scale. Res Nurs Health. 1987 Dec;10(6):357-65. doi: 10.1002/nur.4770100603. PMID 3423307
- [Background] Tiwari R, Kumar R, Malik S, Raj T, Kumar P. Analysis of Heart Rate Variability and Implication of Different Factors on Heart Rate Variability. Curr Cardiol Rev. 2021;17(5):e160721189770. doi: 10.2174/1573403X16999201231203854. PMID 33390146
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Puetz TW. Physical activity and feelings of energy and fatigue: epidemiological evidence. Sports Med. 2006;36(9):767-80. doi: 10.2165/00007256-200636090-00004. PMID 16937952
- [Background] Paluska SA, Schwenk TL. Physical activity and mental health: current concepts. Sports Med. 2000 Mar;29(3):167-80. doi: 10.2165/00007256-200029030-00003. PMID 10739267
- [Background] Rosenbaum S, Tiedemann A, Sherrington C, Curtis J, Ward PB. Physical activity interventions for people with mental illness: a systematic review and meta-analysis. J Clin Psychiatry. 2014 Sep;75(9):964-74. doi: 10.4088/JCP.13r08765. PMID 24813261
- [Background] Mikkelsen K, Stojanovska L, Polenakovic M, Bosevski M, Apostolopoulos V. Exercise and mental health. Maturitas. 2017 Dec;106:48-56. doi: 10.1016/j.maturitas.2017.09.003. Epub 2017 Sep 7. PMID 29150166
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Beser A, Sorjonen K, Wahlberg K, Peterson U, Nygren A, Asberg M. Construction and evaluation of a self rating scale for stress-induced exhaustion disorder, the Karolinska Exhaustion Disorder Scale. Scand J Psychol. 2014 Feb;55(1):72-82. doi: 10.1111/sjop.12088. Epub 2013 Nov 15. PMID 24236500
- [Background] Tanner BA. Validity of global physical and emotional SUDS. Appl Psychophysiol Biofeedback. 2012 Mar;37(1):31-4. doi: 10.1007/s10484-011-9174-x. PMID 22038278
- [Background] Arapovic-Johansson B, Wahlin C, Kwak L, Bjorklund C, Jensen I. Work-related stress assessed by a text message single-item stress question. Occup Med (Lond). 2017 Dec 2;67(8):601-608. doi: 10.1093/occmed/kqx111. PMID 29016877
- [Background] Ensari I, Greenlee TA, Motl RW, Petruzzello SJ. META-ANALYSIS OF ACUTE EXERCISE EFFECTS ON STATE ANXIETY: AN UPDATE OF RANDOMIZED CONTROLLED TRIALS OVER THE PAST 25 YEARS. Depress Anxiety. 2015 Aug;32(8):624-34. doi: 10.1002/da.22370. Epub 2015 Apr 21. PMID 25899389
- [Background] Herring MP, Monroe DC, Gordon BR, Hallgren M, Campbell MJ. Acute Exercise Effects among Young Adults with Analogue Generalized Anxiety Disorder. Med Sci Sports Exerc. 2019 May;51(5):962-969. doi: 10.1249/MSS.0000000000001860. PMID 30531490
- [Background] Loy BD, Cameron MH, O'Connor PJ. Perceived fatigue and energy are independent unipolar states: Supporting evidence. Med Hypotheses. 2018 Apr;113:46-51. doi: 10.1016/j.mehy.2018.02.014. Epub 2018 Feb 19. PMID 29523293
- [Background] McNair D. M., Lorr M., & Droppleman L. Profile of Mood States questionnaire. San Diego (CA): EDITS, 1981.
- [Background] O'Connor PJ. Evaluation of four highly cited energy and fatigue mood measures. J Psychosom Res. 2004 Nov;57(5):435-41. doi: 10.1016/j.jpsychores.2003.12.006. PMID 15581646
- [Background] Sagelv EH, Hopstock LA, Johansson J, Hansen BH, Brage S, Horsch A, Ekelund U, Morseth B. Criterion validity of two physical activity and one sedentary time questionnaire against accelerometry in a large cohort of adults and older adults. BMJ Open Sport Exerc Med. 2020 Feb 26;6(1):e000661. doi: 10.1136/bmjsem-2019-000661. eCollection 2020. PMID 32153981